CLINICAL TRIAL: NCT04910061
Title: A Single-centre Trial to Investigate the Safety and Pharmacokinetics of Orally Administered Nicotinamide Mononucleotide (NMN, 400mg) Over 29 Days of Supplementation in Healthy Adults.
Brief Title: Safety and Pharmacokinetics of Nicotinamide Mononucleotide (NMN) in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seneque SA (Industry)
Collaborators: Dicentra Inc. (Industry); LGD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-NNHSP-01
Record Dates: First submitted 2021-05-10; First posted 2021-06-02 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
Keywords: safety; pharmacokinetics
MeSH Terms: interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Intervention Model Description: A single-arm, non-randomized, non-controlled, monocenter repeated-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMN-C (Experimental): Healthy individuals receiving NMN-C
  Interventions: Dietary Supplement: Nicotinamide mononucleotide (NMN-C)

INTERVENTIONS:
Dietary Supplement: Nicotinamide mononucleotide (NMN-C) — Daily supplementation with NMN-C at 400 mg for 29 days in total

SUMMARY:
The purpose of this study is to investigate the safety, pharmacokinetic profile, and effects of nicotinamide mononucleotide (NMN-C) in healthy adults, 18-65 years of age. The effects will be studied over the course of 30 days in a repeated-dose study through the collection of blood and urine samples, and administration of surveys and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Naturally post-menopausal women with amenorrhea for 1 year will be eligible.
* Females of childbearing potential should be either sexually inactive (abstinent) for 60 days prior to the first dose of the study, throughout the study and for 30 days after completion of the study, or be using an acceptable methods of birth control.
* BMI between 18.5 and 29.9 kg/m2; with a stable weight over the last 3 months (±2 kg).
* Having given written informed consent to participate in the research trial.
* Agrees to maintain current dietary habits and level of physical activity for the trial duration, except as directed by the Nutritionist Agrees to follow dietary guidelines, consume standardized meals, and abide by dietary guidelines for dinner prior to specified visits (as outlined by Nutritionist at screening)

Exclusion Criteria:

* Known or suspected allergy to any of the ingredients in the investigational product or standardized meals.
* Active infection, or history of infection and/or antibiotic use 2 weeks prior to the screening visit as assessed by Investigator.
* Presenting, in the opinion of the Investigator, a clinically significant abnormality with regard to the clinical examination and/or clinical chemistry screening parameters.
* Have a history of, or present with, cardiovascular, renal, hepatic, endocrine, gastrointestinal, or inflammatory disease, as assessed by Investigator.
* Has consumed multivitamins or supplements (such as St. John's Wort) within 1 month prior to the study, or unwilling to discontinue use for the duration of the study
* History of cancer in the last 5 years, or currently has cancer, as assessed by Investigator.
* Has a history of, or current neurological (neurodegenerative diseases, epilepsy) or psychiatric pathology that may impact the participant's ability to comply with the requirements of the protocol, as assessed by Investigator.
* Presenting with immune suppression (e.g. autoimmune disease, HIV), as assessed by Investigator.
* Has undergone surgery in the last 3 months, or has surgery planned during the trial period, as assessed by Investigator.
* Uses concomitant medications including natural health products (excluding contraceptives and PRN or other medications, which in the Investigator's opinion, do not affect the trial outcomes or participant safety).
* Currently following a regimented or restricted diet which in the opinion of the Nutritionist and/or PI would negatively affect the study outcome or participants' ability to comply with study requirements, or has in the 3 months prior to enrollment.
* Plans to change dietary habits and/or activity level during the trial period.
* Frequent consumption of alcohol (> 2 standard servings of alcohol/day on average).
* History of (assessed by PI) or current tobacco use (verified by positive cotinine urinalysis)
* Positive urinalysis for drugs of abuse (amphetamines, Cannabinoids, Cocaine and Opiates)
* Presenting a niacin deficiency, as assessed by Nutritionist's dietary assessment at screening, and Investigator's physical examination.
* Has difficulty swallowing capsules.
* Inability to provide blood and/or urine samples.
* Positive pregnancy test, intent to get pregnant, or breastfeeding.
* Any other condition that, in the opinion of the Investigator, could impair the Investigator's ability to complete the study outcomes and participant safety. Participating simultaneously in another clinical research protocol or having participated in another research study for which the exclusion period would not be completed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Safety as measured by subject incident of treatment-emergent adverse events | between Day 1 and Day 30
  Subject incidence of treatment-emergent adverse events
Safety as measured by subject incident of treatment-emergent clinically significant changes in vital signs | between Day 1 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in vital signs (body temperature, heart rate and blood pressure)
Safety as measured by subject incident of treatment-emergent clinically significant changes in clinical laboratory safety tests. | between Day 1 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete blood count, C reactive protein, AST, ALT, bilirubin, GGT, Alkaline phosphatase, creatinine, creatine kinase, Sodium, Potassium, Chloride)

SECONDARY OUTCOMES:
Change from baseline in NAD+ and NMN concentrations in whole blood | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 1
  NAD+ and NMN will be assessed in blood at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Change from baseline in NAD+ and NMN concentrations in whole blood | Day 1, Day 2, Day 8, Day 15, Day 22, Day 29, Day 30
  NAD+ and NMN will be assessed in blood
Change from baseline in NAD+ metabolites concentrations in plasma | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 1
  MeNAM and NAM will be assessed in plasma at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Change from baseline in NAD+ metabolites concentrations in plasma | Day 1, Day 2, Day 8, Day 15, Day 22, Day 29, Day 30
  MeNAM and NAM will be assessed in plasma
Change from baseline in NAD+ metabolites concentrations in urine | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 1
  MeNAM and Me-2-PY will be assessed in urine at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Change from baseline in NAD+ metabolites concentrations in urine | Day 1, Day 2, Day 8, Day 15, Day 22, Day 29, Day 30
  MeNAM and Me-2-PY will be assessed in urine
Change from baseline in NAD+ and NMN concentrations in whole blood | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 29
  NAD+ and NMN will be assessed in blood at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Change from baseline in NAD+ metabolites concentrations in plasma | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 29
  MeNAM and NAM will be assessed in plasma at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Change from baseline in NAD+ metabolites concentrations in urine | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 hour post-dose on Day 29
  MeNAM and Me-2-PY will be assessed in urine at the following time points : t=0 hours (pre-dose), t=0.25 hours, t=0.5 hours, t=1 hours, t=2 hours, t=4 hours, t=8 hours and t=12 hours after dosing
Changes in body weight | Day 1, Day 29
Tolerance | Day 1, Day 2, Day 8, Day 15, Day 22, Day 29, Day 30
  The number of participants with Adverse Events
Changes in Quality of life | Day 1, Day 29
  the mean changes in the the generic Quality of Life Self-Assessment Questionnaire SF-36 questionnaire score (The SF-36 questionnaire is scaled from a 0 to 100. The lower the score the more disability)
Changes in Sleep quality | Day 1, Day 29
  the mean changes in the Sleep Quality Scale (SQS) score (SQS is providing an overall score ranging from 0 to 84, where lower scores denote a healthier sleep quality)
Changes in Fatigue state | Day 1, Day 29
  the mean changes in the Multidimensional Fatigue Inventory (MFI-20) score (MFI-20 is providing an overall score ranging from 20 to 100 (a higher score indicates a higher level of fatigue).
Change in blood lipid profile from baseline during the intervention period | Day 1, Day 29
  Total cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglyceride concentrations will be evaluated
Change in blood glucose (fasting) from baseline during the intervention period | Day 1, Day 29
  the McNair Cognitive Difficulty Self Questionnaire
Change from baseline in homocysteine concentrations | Day 1, Day 29
  homocysteine level will be evaluated in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Vitalabs Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No